CLINICAL TRIAL: NCT01153464
Title: Effectiveness of Extended Treatment for Drug Dependence - City Supplement
Brief Title: Effectiveness of Extended Treatment for Drug Dependence (ETDD) in the City Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 810106
Record Dates: First submitted 2010-06-24; First posted 2010-06-30 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment As Usual (No Intervention): In this arm, participants are not provided any intervention through the study, they are just followed for research purposes at 3m, 6m, 9m, and 12m post baseline as the comparison group.
- Recovery Support Counseling (Experimental): This group is eligible to receive the telephone based recovery support counseling from paraprofessionals based out of the City of Philadelphia's Department of Behavioral Health.
  Interventions: Behavioral: Recovery Support Counseling

INTERVENTIONS:
Behavioral: Recovery Support Counseling — Telephone based recovery support provided by paraprofessionals at the City of Philadelphia's Behavioral Health Department. Calls are once weekly for 8 weeks, then step down to every other week for the remainder of the year of study participation. Call frequency can be increased as a result of a rise in risk factor/protective factor ratio.
  Arms: Recovery Support Counseling

SUMMARY:
This protocol (a supplement to 805466) is to test whether our telephone continuing care model can be implemented successfully by "real world" publicly funded programs. Participants will be recruited from Philadelphia's Department of Behavioral Health - run drug programs. The investigators will train city telephone care managers to deliver our telephone continuing care intervention to patients in this program. The investigators will randomize 200 to receive this intervention or usual care and follow them for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* (1) qualify for a DSM-IV diagnosis of cocaine dependence, with cocaine use in the 6 months prior to entrance into the City of Philadelphia Department of Behavioral Health facilities or controlled environment;
* (2) 18 to 75 years of age;
* (3) no current psychotic disorder (as assessed with the psychotic screen from the SCID) or evidence of dementia severe enough to prevent participation in outpatient treatment;
* (4) no acute medical problem requiring immediate inpatient treatment;
* (5) no current participation in methadone or other modes of Drug and Alcohol treatment, other than an Intensive Outpatient Program;
* (6) willingness to be randomized and participate in research.
* (7) Finally, because of study follow-up requirements, subjects will be able to provide the name, verified telephone number, and address of at least two contacts who can provide locating information on the patient during follow-up. We will include patients with dependence on other substances, provided that they are cocaine dependent and meet other inclusion criteria.

Exclusion Criteria:

* Current dependence on opiates is an exclusion as those participants may be better served as part of a methadone program rather than a telephone based therapy protocol. Also, if patients are court-ordered to treatment, or otherwise considered prisoners, they will not be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back | 3 month
  abstinence from drug and alcohol use within each 3 month period of the follow-up (as indicated by the TLFB)
Time Line Follow Back | 6 month
  abstinence from drug and alcohol use within each 3 month period of the follow-up (as indicated by the TLFB)
Time Line Follow Back | 9 month
  abstinence from drug and alcohol use within each 3 month period of the follow-up (as indicated by the TLFB)
Time Line Follow Back | 12 month
  abstinence from drug and alcohol use within each 3 month period of the follow-up (as indicated by the TLFB)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States